CLINICAL TRIAL: NCT01105650
Title: Lymphodepleting Chemotherapy and T-Cell Suppression Followed By Allogeneic Natural Killer Cells and IL-2 in Patients With Recurrent Ovarian, Fallopian Tube, Primary Peritoneal Cancer and Advanced Metastatic Breast Cancer (MT2009-30)
Brief Title: Allogeneic Natural Killer (NK) Cells for Ovarian, Fallopian Tube, Peritoneal and Metastatic Breast Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Masonic Cancer Center, University of Minnesota (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2009LS142; MT2009-30 (Other: Blood and Marrow Transplantation Program); 1003M78876 (Other: IRB, University of Minnesota)
Record Dates: First submitted 2010-04-14; First posted 2010-04-16 (Estimated); Results first posted 2017-02-24 (Actual); Last update posted 2017-12-28 (Actual); Status verified 2017-12

CONDITIONS: Ovarian Cancer; Fallopian Tube Cancer; Primary Peritoneal Cancer; Breast Cancer
Keywords: recurrent ovarian cancer; recurrent fallopian tube cancer; recurrent primary peritoneal cancer; refractory ovarian cancer; refractory fallopian tube cancer; refractory peritoneal cancer; metastatic breast cancer
MeSH Terms: conditions — Ovarian Neoplasms; Fallopian Tube Neoplasms; Breast Neoplasms | interventions — fludarabine; fludarabine phosphate; Cyclophosphamide; Cyclosporine; IL32 protein, human; Interleukin-2; Methylprednisolone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Arm 1: CsA (Experimental): Patients receiving Cyclosporine (CsA) and Natural Killer (NK) cells infusion (created from donor lymphapheresis) after preparative regimen of Fludarabine and Cyclophosphamide. Interleukin-2 (IL-2) 6 million units 3 times a week x 6 doses given post NK cell infusion.
  Interventions: Drug: Fludarabine; Drug: Cyclophosphamide; Drug: Cyclosporine; Biological: Natural killer cells; Drug: IL-2; Drug: Interleukin-2
- Arm 2: CsA plus Methylprednisolone (10mg) (Experimental): Patients receiving Cyclosporine (CsA), methylprednisolone and natural killer cells (NK) infusion (created from donor lymphapheresis) after preparative regimen of Fludarabine and Cyclophosphamide. Interleukin-2 (IL-2) 6 million units 3 times a week x 6 doses given post NK cell infusion.
  Interventions: Drug: Fludarabine; Drug: Cyclophosphamide; Drug: Cyclosporine; Biological: Natural killer cells; Drug: IL-2; Drug: Methylprednisolone; Drug: Interleukin-2
- Arm 3: CsA plus Methylprednisolone (1 mg) (Experimental): Patients receiving Cyclosporine (CsA), methylprednisolone and natural killer (NK) cells infusion (created from donor lymphapheresis) after preparative regimen of Fludarabine and Cyclophosphamide. Interleukin-2 (IL-2) 6 million units 3 times a week x 6 doses given post NK cell infusion.
  Interventions: Drug: Fludarabine; Drug: Cyclophosphamide; Drug: Cyclosporine; Biological: Natural killer cells; Drug: IL-2; Drug: Methylprednisolone; Drug: Interleukin-2
- Arm 4: CsA minus Methylprednisolone (Experimental): Patients receiving Cyclosporine (CsA), no methylprednisolone, eliminating IL-2 doses 4-6 and receiving Natural Killer (NK) cells infusion (created from donor lymphapheresis) after preparative regimen of Fludarabine and Cyclophosphamide. Interleukin-2 (IL-2) 6 million units 3 times a week x 3 doses given post NK cell infusion.
  Interventions: Drug: Fludarabine; Drug: Cyclophosphamide; Drug: Cyclosporine; Biological: Natural killer cells; Drug: Interleukin-2

INTERVENTIONS:
Drug: Fludarabine — Administered intravenously, 25 mg/m^2, days -6 through -2 (5 days).
  Other Names: Fludara
Drug: Cyclophosphamide — Administered intravenously, 60 mg/kg, days -5 and -4.
  Other Names: Cytoxan
Drug: Cyclosporine — Administered intravenously, CsA 1.5 mg/kg for target dose range of 150-250 ng/mL day -3 through day +14
  Other Names: Cyclosporine A; CsA
Biological: Natural killer cells — Administered by infusion over less than 1 hour, no more than 8.0 x 10^7 cells/kg will be given.
Drug: IL-2 — Will be given subcutaneously at 9 million units 3 times a week for a total of 6 doses, beginning 4 hours after NK cell infusion. (For patients weighing less than 45 kilograms, will be given at 5 million units/m^2 3 times per week for 6 doses).
  Other Names: Interleukin-2
  Arms: Arm 1: CsA; Arm 2: CsA plus Methylprednisolone (10mg); Arm 3: CsA plus Methylprednisolone (1 mg)
Drug: Methylprednisolone — Administered intravenously (IV) 10 mg/kg Days -2 to +4 and 1 mg/kg Days +5 to +9
  Other Names: Medrol
  Arms: Arm 2: CsA plus Methylprednisolone (10mg); Arm 3: CsA plus Methylprednisolone (1 mg)
Drug: Methylprednisolone — Administered intravenously (IV) 1 mg/kg Days -2 to +9
  Other Names: Medrol
  Arms: Arm 2: CsA plus Methylprednisolone (10mg); Arm 3: CsA plus Methylprednisolone (1 mg)
Drug: Interleukin-2 — Will be given subcutaneously at million units 3 times a week for a total of 3 doses, beginning 4 hours after NK cell infusion. (For patients weighing less than 45 kilograms, will be given at 3 million units/m^2 3 times per week for 6 doses).
  Other Names: IL-2

SUMMARY:
This is a single center phase II trial designed to optimize a clinical platform of lymphodepleting chemotherapy and T-cell suppression to promote the persistence, function, and expansion of allogeneic natural killer (NK) cells in patients with recurrent ovarian, fallopian tube, primary peritoneal cancer and advanced metastatic breast cancer.

DETAILED DESCRIPTION:
The donor NK cells are infused on day 0, after a non-myeloablative preparative regimen of cyclophosphamide and fludarabine plus a cyclosporine A (CsA) based immunosuppressive therapy. Subcutaneous interleukin-2 (IL-2) is started the evening of the NK infusion and continued three times a week for 6 doses total.

Up to 4 sequential immunosuppressive platforms will be tested (Arms 1 and 2 are currently closed) to identify a platform where patients have the potential for successful NK cell expansion (defined as an absolute circulating donor derived NK cell count of > 100 cells/μl 14 days after NK cell infusion). Once a clinical platform is determined, the platform will be expanded to a total of 18 patients. The primary goal of this extended phase is to obtain preliminary efficacy information.

Follow-up for disease response is for 1 year from the NK cell infusion, with the possibility of re-treatment for patients who experience at least a clinical benefit who progress after 6 months.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of recurrent ovarian cancer, fallopian tube, or primary peritoneal cancer that has failed or progressed after at least 2 prior salvage chemotherapy regimens (directed at recurrent/metastatic disease).

OR

* Diagnosis of metastatic breast cancer (female or male) that has progressed on or failed at least one salvage chemotherapy regimen for metastatic disease and that meets the following disease specific related criteria:

  * If estrogen receptor or progesterone receptor positive must have progressed on prior hormonal therapy and/or
  * if HER2-neu positive must have progressed on trastuzumab, lapatinib, or similar agent

Women with a history of both cancers are eligible for this study provided that they currently meet eligibility for one of the diseases. Women who have had another malignancy and have been disease free for at least 3 year, or with a history of completely resected non-melanomatous skin carcinoma or successfully treated in situ carcinoma are eligible.

* Measurable disease per disease specific Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1 - patients with bone as their only site of disease will not be eligible.
* If history of brain metastases must be stable for at least 3 months after treatment - A brain computed tomography (CT) scan will only be required in subjects with known brain metastases at the time of enrollment or in subjects with clinical signs or symptoms suggestive of brain metastases.
* Available related HLA-haploidentical natural killer (NK) cell donor (by at least class I serologic typing at the A&B locus)
* Age 18 years or older
* Karnofsky performance status > or = 50%
* Adequate organ function as determined by the following criteria within 14 days of study enrollment

  * Bone marrow: platelets > or = 80,000 x 10^9/L and hemoglobin > or = 9 g/dL, unsupported by transfusions; absolute neutrophil count (ANC) > or = 1000 x 10^9/L, unsupported by growth colony stimulating factor (G-CSF) or granulocyte-macrophage colony-stimulating factor (GM-CSF)
* Renal function: creatinine (Cr) < or = 2.0 mg/dL
* Liver function: Aspartate aminotransferase (AST), Alanine transaminase (ALT), total bilirubin, alkaline phosphatase < 5 times upper limit of institutional normal (ULN)
* Cardiac: Left ventricular ejection fraction >40% (within 28 days of treatment start)
* Pulmonary function: >50% corrected Carbon Monoxide Diffusing Capacity (DLCO) and Forced Expiratory Volume in One Second (FEV1), if presence of pleural effusion due to metastatic disease >40% corrected DLCO and FEV1 is acceptable (within 28 days of treatment start)
* Able to be off prednisone or other immunosuppressive medications for at least 3 days prior to Day 0
* At least 14 days must lapse between last prior anti-cancer treatment and 1st day of preparative regimen
* Voluntary written informed consent

Exclusion Criteria:

* Pregnant or nursing - The agents used in this study may be teratogenic to a fetus and there is no information on the excretion of agents into breast milk. Participants of childbearing potential must have a blood test or urine study within 14 days prior to registration to rule out pregnancy and agree to use adequate birth control during study treatment
* Active infection - subjects must be afebrile, off antibiotics, and with no uninvestigated radiologic lesions (infiltrates or lesions with negative cultures or biopsies) are allowed

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2010-07; Primary Completion 2014-04 (Actual); Study Completion 2014-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Melissa Geller, MD, Principal Investigator — Masonic Cancer Center, University of Minnesota
Locations (1):
- Masonic Cancer Center, University of Minnesota, Minneapolis, Minnesota, United States

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Up to 4 sequential immunosuppressive platforms (study arms) were tested to identify a platform where patients have the potential for successful Natural Killer (NK) cell expansion (defined as an absolute circulating donor derived NK cell count of > 100 cells/μl 14 days after NK cell infusion).
Groups:
- Arm 1: CsA: Fludarabine: Administered intravenously, 25 mg/m^2, days -6 through -2 (5 days).
  Cyclophosphamide: Administered intravenously, 60 mg/kg, days -5 and -4.
  Cyclosporine (CsA): Administered intravenously, 1.5 mg/kg for target dose range of 150-250 ng/mL day -3 through day +14
  Natural Killer cells: Administered by infusion over less than 1 hour; no more than 8.0 x 10^7 cells/kg will be given.
  Interleukin- 2 (IL-2): Given subcutaneously at 9 million units 3 times a week for a total of 6 doses, beginning 4 hours after NK cell infusion. (For patients weighing less than 45 kilograms, IL-2 will be given at 5 million units/m^2 3 times per week for 6 doses).
- Arm 2: CsA/Methylprednisolone (10mg)/6 Doses of Interleukin-2: Fludarabine: Administered intravenously, 25 mg/m^2, days -6 through -2 (5 days).
  Cyclophosphamide: Administered intravenously, 60 mg/kg, days -5 and -4.
  Cyclosporine (CsA): Administered intravenously, 1.5 mg/kg for target dose range of 150-250 ng/mL day -3 through day +14
  Natural Killer cells: Administered by infusion over less than 1 hour; no more than 8.0 x 10^7 cells/kg will be given.
  Interleukin- 2 (IL-2): Given subcutaneously at 9 million units 3 times a week for a total of 6 doses, beginning 4 hours after NK cell infusion. (For patients weighing less than 45 kilograms, IL-2 will be given at 5 million units/m^2 3 times per week for 6 doses).
  Methylprednisolone: Administered intravenously,10 mg/kg Days -2 to +4 and 1 mg/kg Days +5 to +9.
- Arm 3: CsA/Methylprednisolone (1mg)/6 Doses of Interleukin-2: Fludarabine: Administered intravenously, 25 mg/m^2, days -6 through -2 (5 days).
  Cyclophosphamide: Administered intravenously, 60 mg/kg, days -5 and -4.
  Cyclosporine (CsA ): Administered intravenously, 1.5 mg/kg for target dose range of 150-250 ng/mL day -3 through day +14
  Natural Killer cells: Administered by infusion over less than 1 hour; no more than 8.0 x 10^7 cells/kg will be given.
  Interleukin- 2 (IL-2): Given subcutaneously at 9 million units 3 times a week for a total of 6 doses, beginning 4 hours after NK cell infusion. (For patients weighing less than 45 kilograms, IL-2 will be given at 5 million units/m^2 3 times per week for 6 doses).
  Methylprednisolone: Administered intravenously, 1 mg/kg Days -2 to +9
- Arm 4: CsA/no Methylprednisolone/3 Doses of Interleukin-2: Fludarabine: Administered intravenously, 25 mg/m^2, days -6 through -2 (5 days).
  Cyclophosphamide: Administered intravenously, 60 mg/kg, days -5 and -4.
  Cyclosporine (CsA ): Administered intravenously, 1.5 mg/kg for target dose range of 150-250 ng/mL day -3 through day +14
  Natural Killer cells: Administered by infusion over less than 1 hour; no more than 8.0 x 10^7 cells/kg will be given.
  Interleukin-2 (IL-2): Given subcutaneously at 9 million units 3 times a week for a total of 3 doses, beginning 4 hours after NK cell infusion. (For patients weighing less than 45 kilograms, IL-2 will be given at 3 million units/m^2 3 times per week for 3 doses).
Period: Overall Study
Arm/Group | Arm 1: CsA | Arm 2: CsA/Methylprednisolone (10mg)/6 Doses of Interleukin-2 | Arm 3: CsA/Methylprednisolone (1mg)/6 Doses of Interleukin-2 | Arm 4: CsA/no Methylprednisolone/3 Doses of Interleukin-2
Started | 3 | 3 | 7 | 0 (Arm 3 was determined to be successful, thus eliminating the need to test Arm 4.)
Completed | 3 | 3 | 7 | 0
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm 1: CsA | Arm 2: CsA/Methylprednisolone (10mg)/6 Doses of Interleukin-2 | Arm 3: CsA/Methylprednisolone (1mg)/6 Doses of Interleukin-2 | Total
Number analyzed (Participants) | 3 | 3 | 7 | 13
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 0 | 2 | 5 | 7
  >=65 years | 3 | 1 | 2 | 6
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 3 | 7 | 13
  Male | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Response Rate
Description: Response includes Complete Response (CR), Partial Response (PR), and Stable Disease (SD) as defined by Response Evaluation Criteria In Solid Tumors Criteria (RECIST v.1.1) for target lesions and assessed by CT or MRI. Complete Response (CR), disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions; Stable Disease (SD), neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for Progressive Disease.
Time Frame: Month 3
Measure: Number; unit: participants
Arm/Group | Arm 1: CsA | Arm 2: CsA/Methylprednisolone (10mg)/6 Doses of Interleukin-2 | Arm 3: CsA/Methylprednisolone (1mg)/6 Doses of Interleukin-2
Number analyzed (Participants) | 3 | 3 | 7
participants | 1 | 2 | 4

2. Secondary Outcome: Time to Disease Progression
Description: Time from study entry until progressive disease or data collection cutoff.
Time Frame: 1 Year
Population: Number of participants with progressive disease at one year:
  Arm 1: 2 out of 3; Arm 2: 1 out of 3; Arm 3: 5 out of 7
Measure: Median (Full Range); unit: days
Arm/Group | Arm 1: CsA | Arm 2: CsA/Methylprednisolone (10mg)/6 Doses of Interleukin-2 | Arm 3: CsA/Methylprednisolone (1mg)/6 Doses of Interleukin-2
Number analyzed (Participants) | 3 | 3 | 7
days | 52 [28 to 76] | 98 [98 to 98] | 100 [94 to 201]

3. Secondary Outcome: Number of Participants With Progressive Disease at One Year
Time Frame: 1 Year
Measure: Count of Participants; unit: Participants
Arm/Group | Arm 1: CsA | Arm 2: CsA/Methylprednisolone (10mg)/6 Doses of Interleukin-2 | Arm 3: CsA/Methylprednisolone (1mg)/6 Doses of Interleukin-2
Number analyzed (Participants) | 3 | 3 | 7
Participants | 2 | 1 | 5

4. Secondary Outcome: Overall Survival
Description: Number of participants alive at 1 year.
Time Frame: 1 Year
Measure: Number; unit: participants
Arm/Group | Arm 1: CsA | Arm 2: CsA/Methylprednisolone (10mg)/6 Doses of Interleukin-2 | Arm 3: CsA/Methylprednisolone (1mg)/6 Doses of Interleukin-2
Number analyzed (Participants) | 3 | 3 | 7
participants | 0 | 1 | 3

ADVERSE EVENTS:
Arm/Group | Arm 1: CsA | Arm 2: CsA/Methylprednisolone (10mg)/6 Doses of Interleukin-2 | Arm 3: CsA/Methylprednisolone (1mg)/6 Doses of Interleukin-2
Serious Adverse Events (participants affected / at risk) | 3/3 | 3/3 | 5/7
Other Adverse Events (participants affected / at risk) | 3/3 | 3/3 | 7/7
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Arm 1: CsA (N=3) | Arm 2: CsA/Methylprednisolone (10mg)/6 Doses of Interleukin-2 (N=3) | Arm 3: CsA/Methylprednisolone (1mg)/6 Doses of Interleukin-2 (N=7)
Abdominal pain (Gastrointestinal disorders) | 1 | 0 | 0
Death NOS (General disorders) | 3 | 2 | 1
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Hearing impairmed (Ear and labyrinth disorders) | 0 | 1 | 0
Vestibular disorder (Ear and labyrinth disorders) | 0 | 1 | 0
Blurred vision (Eye disorders) | 0 | 1 | 0
Acute kidney injury (Renal and urinary disorders) | 0 | 1 | 1
Hypertension (Vascular disorders) | 0 | 1 | 0
Atrial flutter (Cardiac disorders) | 0 | 0 | 1
Fever (General disorders) | 0 | 0 | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Arm 1: CsA (N=3) | Arm 2: CsA/Methylprednisolone (10mg)/6 Doses of Interleukin-2 (N=3) | Arm 3: CsA/Methylprednisolone (1mg)/6 Doses of Interleukin-2 (N=7)
Acute kidney injury (Renal and urinary disorders) | 1 | 1 | 1
Ascites (Gastrointestinal disorders) | 2 | 1 | 0
Capillary leak syndrome (Vascular disorders) | 2 | 0 | 3
Chills (General disorders) | 3 | 3 | 7
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 3 | 3 | 5
Edema (General disorders) | 2 | 3 | 5
Fever (General disorders) | 3 | 2 | 6
Headache (Nervous system disorders) | 1 | 1 | 4
Hypertension (Vascular disorders) | 3 | 2 | 7
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 3 | 2 | 4
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 0
Rash/Desquamation (Skin and subcutaneous tissue disorders) | 2 | 1 | 2
Infusion related reaction (General disorders) | 2 | 0 | 3
Injection Site Reaction (General disorders) | 1 | 0 | 5
Neutropenic fever (Blood and lymphatic system disorders) | 1 | 3 | 6
Pneumonitis/Pulmonary Infiltrates (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1
Depressed level of consciousness (Nervous system disorders) | 0 | 1 | 0
Hallucinations (Nervous system disorders) | 0 | 1 | 0
Hypotension (Vascular disorders) | 0 | 2 | 3
Dizziness (Nervous system disorders) | 0 | 1 | 0
Hearing loss (Ear and labyrinth disorders) | 0 | 1 | 0
Atrial fibrillation (Cardiac disorders) | 0 | 1 | 0
Confusion/Disoriented (Nervous system disorders) | 0 | 1 | 0
Double vision (Eye disorders) | 0 | 1 | 0
Foot pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Strange dreams (Nervous system disorders) | 0 | 1 | 0
Creatinine Increased (Investigations) | 0 | 0 | 4
Hypokalemia (Metabolism and nutrition disorders) | 0 | 0 | 1
Body aches (General disorders) | 0 | 0 | 2
Night sweats (General disorders) | 0 | 0 | 1
Weight gain (Investigations) | 0 | 0 | 3
Fall (Injury, poisoning and procedural complications) | 0 | 0 | 1
Nausea (Gastrointestinal disorders) | 0 | 0 | 1
Pain with stools (Gastrointestinal disorders) | 0 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No